CLINICAL TRIAL: NCT05015413
Title: Effect of Shockwave Versus Low Level Laser Therapy on Sacroiliac Joint Pain in Postnatal Women
Brief Title: Effect of Shockwave Versus LLL Therapy on Sacroiliac Joint Pain in Postnatal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samar Mimi Mohamed Okby (Other)
Responsible Party: Sponsor-Investigator, Samar Mimi Mohamed Okby, Physical therapist in al Agoza police hospital, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012/003237
Record Dates: First submitted 2021-07-14; First posted 2021-08-20 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Sacroiliac Joint Pain

STUDY DESIGN:
Intervention Model Description: Group A will receive shock wave therapy Group B will receive low level laser therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shock wave group (Experimental): Group A will receive shockwave therapy 2 session per week for 6 weeks
  Interventions: Device: Shockwave
- low level laser group (Experimental): Group B will receive low level laser therapy 2 session per week for 6 weeks
  Interventions: Device: Shockwave

INTERVENTIONS:
Device: Shockwave — Shock wave master 500 Germany

SUMMARY:
Sacroiliac joint pain is the most causes of back pain In pregnancy caused ligament laxity in sacroiliac joint so cause pain and this pain continue after natal Shock wave is new conservative treatment used in physical therapy Shock wave is most effective for sacroiliac joint pain Low level laser is a most effective pain relive and effective on sacroiliac joint pain

DETAILED DESCRIPTION:
The study is to determine if there is any difference between the effect of shockwave and low level laser therapy on sacroiliac joint pain in postnatal women This study will be randomly distributed into two equal group Group A consisted of 25 postpartum women complaining from sacroiliac joint pain . They will receive shockwave therapy 2 session per week for 6 weeks Group B consisted of 25 postpartum women complaining from sacroiliac joint pain . They will receive low level laser therapy 2 session per week for 6 weeks

Evaluation procedures History taking recording in recording data sheet Weight and height measurement by calculate BMI Disability assessment by OWDI Pain assessment by VAS scale Assessment of pressure of pain threshold by pressure algometry

ELIGIBILITY:
Inclusion Criteria:

* postnatal women suffering from sacroiliac joint pain for at least 3 months.
* They should have moderate to severe pain .
* They should have positive findings in at least 3 of 5 provocation sacroiliac joint tests

Exclusion Criteria:

* lumber or hip joint pathology
* Acute pelvic bacterial or viral infection .
* Receiving corticosteroid injections within the previous 6 weeks

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postnatal women
Enrollment: 50 (Estimated)
Dates: Start 2021-11-25 (Estimated); Primary Completion 2021-12-03 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
Sacroiliac joint pain | About two months
  •Pain intensity: it will by measure by VAS it's presented as 10 cm horizontal line on which the patient pain intensity is point between no pain at zero score to extreme pain at 10 score .
Functional disability | About 2 month
  •Functional disability :it will be measure by oswestry disability index it is 10 point Patient reported outcome questionnaire which the higher score mean its the worst and the low score mean its the better outcome.
Pain pressure threshold | About 2 month
  •Pain pressure threshold : it will be measure by a device Called pressure algometry

IPD SHARING:
Plan to Share IPD: Yes